CLINICAL TRIAL: NCT06408038
Title: Are CK+/CD45+ Double-Positive Circulating Cells of Tumor-origin? Characterization in METAstatic Breast Cancer
Acronym: DP METABREAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Collaborators: Fondation Toulouse Cancer Santé (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 24SEIN02
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic Breast Cancer; CK+/CD45+; Double-Positive circulating cells
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with MBC (Other)
  Interventions: Other: For each patient included, the samples described below will be collected:

INTERVENTIONS:
Other: For each patient included, the samples described below will be collected: — * A single blood sample will be taken before initiation of the metastatic treatment line. The volume of total blood sampled is 34mL.
  * A tumour sample (FFPE block already archived) from a metastasis (other than bone) if available or, failing this, from the primary breast tumour, will be sent to the sponsor in order to meet the objectives of the study.
  Once the blood sample has been taken, patients will have completed their participation in the study.

SUMMARY:
A prospective, single-centre, proof-of-concept pilot study in patients with metastatic breast cancers (MBC) (whatever the immunohistochemical subtype) treated at the IUCT-O. Eligible patients will be selected and informed of this study during a medical consultation for cancer that has metastasised, has relapsed or is progressing metastatically, by medical oncologists at the Oncopole Claudius Regaud (OCR). Then, with the patient's agreement and before the start of anti-tumour treatment, a blood sample will be taken to detect DP-circulating cells. A breast cancer tumour sample (non-bone metastasis or, failing that, primary tumour) must be available (FFPE archived tumour block).

Each patient will participate in the study for one day.

60 patients will be included in this interventional study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with metastatic breast cancer eligible for 1st, 2nd or 3rd line treatment at stage IV, regardless of immunohistochemical subtype (triple-negative, RH+/HER2-negative or HER2-positive).
2. Patient with metastatic disease or metastatic relapse or progression who has not yet started 1st line treatment for metastatic disease or line 2 or line 3.
3. Tumour sample available (archived tumour block): non-bone metastasis preferred if available or, failing this, primary breast tumour.
4. Age ≥ 18 years and WHO ≤ 2.
5. Patient affiliated to a French Social Security scheme.
6. Patient having signed his/her informed consent prior to inclusion in the study and prior to any specific procedure for the study.

Exclusion Criteria:

1. Associated pathology(ies) likely to prevent the study procedure from running smoothly.
2. Any psychological, family, geographical or sociological condition that prevents compliance with the medical monitoring and/or procedures set out in the study protocol.
3. Patient who has forfeited his/her freedom by administrative or legal award or who is under legal protection (curatorship and guardianship, protection of justice).
4. Patient who has presented with another solid tumour (excluding carcinoma in situ of the breast or cervix) within 5 years.
5. Pregnant patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-06-25 (Actual); Primary Completion 2025-10-08 (Actual); Study Completion 2025-10-08 (Actual)

PRIMARY OUTCOMES:
Rate of patients with proven tumour origin of DP-circulating cells. This is defined as the number of patients with proven tumour origin of DP-circulating cells out of the number of patients with DP-circulating cells. | Approximately 16 months after the start of the study

SECONDARY OUTCOMES:
The presence and number of DP-circulating cells and conventional circulating tumor cells (CTCs). | Approximately 16 months after the start of the study
  The heterogeneity of DP-circulating cells will be estimated by the penetrance of genomic alterations in a given patient, which will give us information on the sub-clonality of the alteration (shared by x percent of cells), but also by single cell DNA sequencing (scDNAseq).

CONTACTS AND LOCATIONS:
Locations (1):
- IUCT-O, Toulouse, France